CLINICAL TRIAL: NCT00946530
Title: Light Treatment for Sleep/Wake Disturbances in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Jerome A Yesavage,, Professor of Psychiatry, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-06302009-2840; 1677 (Other: Stanford University IRB)
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Light (Experimental): received bright light
  Interventions: Device: Bright light
- Control (Placebo Comparator): received regular light
  Interventions: Device: Control

INTERVENTIONS:
Device: Bright light — Participants uses bright light
  Arms: Bright Light
Device: Control — Participants uses dim light
  Arms: Control

SUMMARY:
The aim of this study is to demonstrate the efficacy of timed exposure to bright light for the treatment of disturbed nighttime sleep and daytime wake in community-dwelling dementia patients and their caregivers, and to determine if there are genetic relationships between memory problems and sleep problems

DETAILED DESCRIPTION:
1. Efficacy: Up to 4 weeks of morning bright light exposure will be more efficacious than morning dim light in consolidating nighttime sleep as assessed by actigraphy.
2. Predictors of response: We expect the primary predictor of treatment response will be initial MMSE score. Secondary predictors include baseline sleep/wake and circadian parameters and age.
3. Effectiveness: Bright light treatment will be more effective than dim light in improving quality of life.
4. An understanding of some of the genetic markers of memory and/or sleep problems.

ELIGIBILITY:
Inclusion Criteria:Alzheimer's Disease Patients:

* Stanford Alzheimer's Disease Core Center member or potential member, with diagnostic criteria met for probable AD, living with caregiver willing to participate in the protocol
* Non-institutionalized

Caregivers:

* Living in home of AD patient and willing to participate in protocol Exclusion Criteria:Alzheimer's Disease Patients:
* History of manic or bipolar disorder
* Prior bright light treatment
* Irregular or non-24 hour sleep/wake cycle
* Positive result on multi-staged RLS/PLMD
* Medical/Ophthalmologic Exclusions
* RDI >20 on overnight EdenTrace® recording

Caregivers:

* History of manic or bipolar disorder
* Medical/Ophthalmologic Exclusions

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Yesavage, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
This was not required at the time.

REFERENCES:
- [Result] Spira AP, Friedman L, Beaudreau SA, Ancoli-Israel S, Hernandez B, Sheikh J, Yesavage J. Sleep and physical functioning in family caregivers of older adults with memory impairment. Int Psychogeriatr. 2010 Mar;22(2):306-11. doi: 10.1017/S1041610209991153. Epub 2009 Nov 30. PMID 19943990
- [Result] Friedman L, Spira AP, Hernandez B, Mather C, Sheikh J, Ancoli-Israel S, Yesavage JA, Zeitzer JM. Brief morning light treatment for sleep/wake disturbances in older memory-impaired individuals and their caregivers. Sleep Med. 2012 May;13(5):546-9. doi: 10.1016/j.sleep.2011.11.013. Epub 2012 Mar 10. PMID 22406033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community, from 2004-2008
Pre-assignment Details: diagnosis changed for 2 care-recipients, so 2 dyads were not included in the final analysis.
Groups:
- Bright Light - AD Patient: AD Participants received bright light for 30 minutes every day within 30 minutes of arising for 2 weeks
- Dim Light (Control) - AD Patients: AD Participants received dim light for 30 minutes every day within 30 minutes of arising for 2 weeks
- Bright Light - Caregiver: Caregiver Participants received bright light for 30 minutes every day within 30 minutes of arising for 2 weeks
- Dim Light (Control) - Caregiver: Caregiver Participants received dim light for 30 minutes every day within 30 minutes of arising for 2 weeks
Period: Overall Study
Arm/Group | Bright Light - AD Patient | Dim Light (Control) - AD Patients | Bright Light - Caregiver | Dim Light (Control) - Caregiver
Started | 32 (32 dyads consisting of 1 AD patient and 1 caregiver were assigned the Bright Light Arm) | 27 (27 dyads consisting of 1 AD patient and 1 caregiver were assigned to the Dim Light (Control) arm) | 32 (32 dyads consisting of 1 AD patient and 1 caregiver were assigned the Bright Light Arm) | 27 (27 dyads consisting of 1 AD patient and 1 caregiver were assigned to the Dim Light (Control) arm)
Completed | 31 (31 dyads consisting of 1 AD patient and 1 caregiver completed the Bright Light Arm) | 23 (23 dyads consisting of 1 AD patient and 1 caregiver completed to the Dim Light (Control) arm) | 31 (31 dyads consisting of 1 AD patient and 1 caregiver completed the Bright Light Arm) | 23 (23 dyads consisting of 1 AD patient and 1 caregiver were assigned to the Dim Light (Control) arm)
Not Completed | 1 | 4 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 3
Not completed — Physician Decision | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Memory impaired older adults and their caregivers
Groups:
- Bright Light-AD Patients: AD patients received bright light
- Dim Light (Control) - AD Patients: AD patients received dim light in the Control condition
- Bright Light - Caregivers: Caregivers received bright light
- Dim Light (Control) - Caregivers: Caregivers received dim light in the Control condition
- Total: Total of all reporting groups
Arm/Group | Bright Light-AD Patients | Dim Light (Control) - AD Patients | Bright Light - Caregivers | Dim Light (Control) - Caregivers | Total
Number analyzed (Participants) | 31 | 23 | 31 | 23 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 31 | 23 | 31 | 23 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 22 | 14 | 59
  Male | 19 | 12 | 9 | 9 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 5 | 0 | 8
  Not Hispanic or Latino | 28 | 23 | 26 | 23 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 29 | 22 | 29 | 22 | 102
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 23 | 31 | 23 | 108

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time
Description: The amount of actual sleep time in a sleep episode.
Time Frame: 2 weeks
Population: dyads consisting of 1 AD patient and 1 caregiver
Measure: Mean (Standard Deviation); unit: units on a scale (minutes)
Groups:
- Bright Light - AD Patient: AD patient received bright light
- Dim Light (Control) - AD Patients: AD patient received regular (dim) light
- Bright Light - Caregiver: Caregiver received Bright Light
- Dim Light (Control) - Caregiver: Caregiver received regular (dim) Light
Arm/Group | Bright Light - AD Patient | Dim Light (Control) - AD Patients | Bright Light - Caregiver | Dim Light (Control) - Caregiver
Number analyzed (Participants) | 31 | 23 | 31 | 23
units on a scale (minutes) | 393 (127) | 420 (125) | 398 (65.4) | 409 (84.9)

2. Secondary Outcome: WASO (Wake After Sleep Onset)
Description: WASO (Wake After Sleep Onset): the amount of time test subjects have spent awake after initially falling sleep and before they awaken for good.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (minutes)
Arm/Group | Bright Light - AD Patient | Dim Light (Control) - AD Patients | Bright Light - Caregiver | Dim Light (Control) - Caregiver
Number analyzed (Participants) | 31 | 23 | 31 | 23
units on a scale (minutes) | 124 (111) | 107 (110) | 63.4 (60.0) | 61.0 (64.8)

ADVERSE EVENTS:
Time Frame: 5 years
Description: No serious adverse events.
Arm/Group | Bright Light-AD Patients | Dim Light (Control) - AD Patients | Bright Light - Caregivers | Dim Light (Control) - Caregivers
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/27 | 0/32 | 0/27
Other Adverse Events (participants affected / at risk) | 0/32 | 0/27 | 0/32 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes